CLINICAL TRIAL: NCT02659241
Title: A Pilot Study of Wee1 Inhibition Induction Prior to Tumor Reductive Surgery in Ovarian Cancer
Brief Title: Adavosertib Before Surgery in Treating Patients With Advanced High Grade Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0519; NCI-2016-00118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0519 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Fallopian Tube Carcinoma; Advanced Ovarian Carcinoma; Advanced Primary Peritoneal Carcinoma; Carcinomatosis; Fallopian Tube High Grade Serous Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Carcinoma; Fallopian Tube Neoplasms | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (adavosertib) (Experimental): Patients receive adavosertib PO QD on days 1-5. Patients then undergo standard of care laparoscopy. Patients may also receive adavosertib PO QD on days 8-12, 15-19, and 22-26 for up to 28 days based on surgery schedule.
  Interventions: Drug: Adavosertib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot early phase I trial studies how adavosertib affects the tumor deoxyribonucleic acid (DNA) of patients undergoing surgery for high grade (fast growing or aggressive) ovarian, fallopian tube, or primary peritoneal cancer that has spread to other places in the body (advanced). Certain characteristics in the DNA of these patients may affect how well they respond to treatment. Learning how adavosertib affects DNA in tumor cells may help doctors plan effective treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To explore baseline levels and effects of adavosertib (AZD1775) on DNA copy number, mutation, and level of ribonucleic acid (RNA) and protein expression (together described as "molecular results") in tumor protein p53 (p53)-related pathways before and after treatment in women with primary advanced high grade serous ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. To correlate molecular results to clinical endpoints including response and survival.

II. To correlate molecular results to pathologic endpoints including tumor volume and apoptosis.

III. To compare DNA copy number and level of RNA and protein expression in p53-related pathways in tissue from patients treated with AZD1775 to those untreated with AZD1775 in the preoperative period.

IV. To determine the toxicity of AZD1775 given preoperatively, with a focus on postoperative wound healing.

V. To determine the feasibility of treating preoperatively with AZD1775.

OUTLINE:

Patients receive adavosertib orally (PO) once daily (QD) on days 1-5. Patients then undergo standard of care laparoscopy. Patients may also receive adavosertib PO QD on days 8-12, 15-19, and 22-26 for up to 28 days based on surgery schedule.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with presumed advanced-stage high grade serous ovarian, fallopian tube, or primary peritoneal carcinoma, based on the presence of carcinomatosis, and/or elevated cancer antigen (CA)125, and/or ovarian mass(es), or at the discretion of the treating physician
* Medically able to undergo primary cytoreductive surgery, at least 13 days and up to 28 days after starting study drug, as determined by treating physician
* No prior therapy for high-grade serous ovarian, fallopian tube, or primary peritoneal carcinoma
* Patients must be able to swallow and tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of AZD1775 (e.g. uncontrolled nausea, vomiting, or diarrhea; malabsorption syndrome; ulcerative disease); Note: patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN)
* Absolute neutrophil count >= 1,500/mcL (within 7 days prior to initiation of therapy)
* Hemoglobin >= 9 gm/dL (within 7 days prior to initiation of therapy)
* Platelets >= 100,000/mcL (within 7 days prior to initiation of therapy)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 7 days prior to initiation of therapy)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal unless the liver is involved with tumor, in that case, AST and ALT must be =< 5 x upper limit of normal (within 7 days prior to initiation of therapy)
* Creatinine clearance > 50 mL/min (assessed by Cockcroft Gault estimation) and creatinine < 1.5 x ULN (within 7 days prior to initiation of therapy)
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Women of childbearing potential (WoCBP) may be included only if acceptable contraception is in place for two weeks before study entry, for the duration of the study and for 90 days after the last dose of AZD1775; WoCBP are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause); acceptable methods of contraception include true abstinence in line with the preferred and usual lifestyle choice of the patient, tubal ligation, vasectomized partner, barrier methods (eg, cap plus spermicide, sponge plus spermicide, diaphragm plus spermicide, or male condom plus a spermicide), intrauterine device methods (eg, Copper T or Levonorgestrel-releasing intrauterine system), or hormonal methods (eg, any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent and that is administered via the oral, subcutaneous, transdermal, intrauterine, or intramuscular route as an implant, hormone shot or injection, combined pill, minipill or patch); all methods of contraception (with the exception of total abstinence) should be used in combination with the use of a condom by their male sexual partner for intercourse; periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control; all WoCBP must have a negative pregnancy test within 3 days prior to study the initiation of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women must not breast-feed while taking the study medications
* Patients must be able to understand and willing to sign an informed consent

Exclusion Criteria:

* Prior treatment for ovarian, fallopian tube, or primary peritoneal cancer
* Current receipt of any other investigational agents or any additional anti-cancer agents for this or any other disease
* Known central nervous system (CNS) disease other than neurologically stable, treated brain metastases -- defined as metastasis having no evidence of progression or hemorrhage after treatment for at least 2 weeks
* Presence of other active cancers; patients with stage I cancer who have received definitive local treatment within the last 3 years, and whom are considered unlikely to recur, are eligible; all patients with previously treated in-situ carcinoma (i.e., non-invasive) are eligible, as are patients with prior non-melanoma skin cancers
* Major surgical procedures =< 28 days of beginning study treatment, or minor surgical procedures =< 7 days (minor procedures done at time of laparoscopy are allowed); no waiting required following port-a-cath placement
* Significant symptom burden from presumed diagnosis including large volume ascites, pain requiring narcotic medication, or shortness of breath on exertion
* Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Corrected QT interval (QTc) > 470 msec (as calculated by Fridericia correction formula) at study entry or congenital long QT syndrome
* Caution should be exercised when inhibitors or substrates of P-glycoprotein (P-gP), substrates of cytochrome P450 family 1 subfamily A member 2 (CYP1A2) with a narrow therapeutic range, sensitive substrates of cytochrome P450 family 2 subfamily C member 19 (CYP2C19) or CYP2C19 substrates with a narrow therapeutic range are administered with AZD1775
* Herbal preparations are not allowed throughout the study; these herbal medications include, but are not limited to: St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng; not willing to avoid grapefruit, grapefruit juices, grapefruit hybrids, Seville oranges, pummelos, and exotic citrus fruits from 14 days prior to the dose of study medication and during the entire study due to potential CYP3A4 interaction with the study medication; orange juice is allowed
* Any known hypersensitivity or contraindication to the components of study treatment
* Pregnant or breast-feeding
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases (e.g., severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease], uncontrolled chronic renal diseases [glomerulonephritis, nephritic syndrome, Fanconi syndrome or renal tubular acidosis]), serious active infection or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension (blood pressure >= 140/90), active bleeding diatheses or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus; screening for chronic conditions and infectious diseases is not required
* As judged by the investigator, the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements
* Subject has had prescription or non-prescription drugs or other products known to be sensitive cytochrome P450 family 3 subfamily A member 4 (CYP3A4) substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors / inducers of CYP3A4 which cannot be discontinued two weeks prior to day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug; co-administration of aprepitant or fosaprepitant during this study is prohibited
* AZD1775 is an inhibitor of breast cancer resistance protein (BCRP).; the use of statins including atorvastatin are prohibited and patients should be moved on to non-breast cancer resistance protein (BCRP) alternatives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in level of deoxyribonucleic acid (DNA) copy number in p53-related pathways | Baseline up to 28 days
  Descriptive statistics and graphical methods will be used to summarize the change in DNA copy number from pre-treatment to post-treatment with adavosertib. These changes for untreated patients will also be summarized. A paired t-test will be used to test that mean changes from pre-treatment to post-treatment are different from 0 if the changes are found to be normally distributed. Otherwise, median changes from pre-treatment to post-treatment will be tested with a Wilcoxon signed-rank test. A 2-sample t-test will be used to compare mean changes between treated and untreated patients if the changes are normally distributed. Otherwise, median changes will be compared between treated and untreated patients with a Wilcoxon rank sum test.
Change in level of mutation in p53-related pathways | Baseline up to 28 days
Change in level of ribonucleic acid (RNA) expression in p53-related pathways | Baseline up to 28 days
  Descriptive statistics and graphical methods will be used to summarize the change in RNA protein expression from pre-treatment to post-treatment with adavosertib. These changes for untreated patients will also be summarized. A paired t-test will be used to test that mean changes from pre-treatment to post-treatment are different from 0 if the changes are found to be normally distributed. Otherwise, median changes from pre-treatment to post-treatment will be tested with a Wilcoxon signed-rank test. A 2-sample t-test will be used to compare mean changes between treated and untreated patients if the changes are normally distributed. Otherwise, median changes will be compared between treated and untreated patients with a Wilcoxon rank sum test. RNA protein expression will also be determined as present/absent. An exact binomial test will be used to assess the proportion of patients treated with adavosertib that exhibit an increase (or decrease) in RNA protein expression greater than 50%.
Change in level of protein expression in p53-related pathways | Baseline up to 28 days
  McNemar's test will be used to compare changes based on protein expression results. Fisher's exact test will be used to compare protein expression results between treated and untreated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - MD Anderson in The Woodlands, Conroe, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- [Derived] Sun C, Fang Y, Labrie M, Li X, Mills GB. Systems approach to rational combination therapy: PARP inhibitors. Biochem Soc Trans. 2020 Jun 30;48(3):1101-1108. doi: 10.1042/BST20191092. PMID 32379297
- See also: MD Anderson Cancer Center — http://www.mdanderson.org